CLINICAL TRIAL: NCT06740214
Title: Analgesic Efficacy of Different Liposomal Bupivacaine Doses in the Adductor Canal Block for Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Analgesic Efficacy of Different Liposomal Bupivacaine Doses in the Adductor Canal Block for Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW24-691
Record Dates: First submitted 2024-11-29; First posted 2024-12-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative; Analgesic Effect; Total Knee Arthroplasty; Liposomal Bupivacaine; Dose Response Relationship, Drug
Keywords: adductor canal block; local infiltration analgesia; liposomal bupivacaine; opioid consumption; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACB using 20ml 0.5% standard bupivacaine (SB-ACB) (Active Comparator): adductor canal block with 20ml 0.5% standard bupivacaine only
  Interventions: Drug: 0.5% standard bupivacaine only
- ACB using 10ml 1.33% liposomal bupivacaine with 10 ml 0.5% standard bupivacaine (LB10-ACB) (Experimental): adductor canal block with 10ml 1.33% liposomal bupivacaine (133mg) plus 10ml 0.5% standard bupivacaine
  Interventions: Drug: 1.33% liposomal bupivacaine with 0.5% standard bupivacaine
- ACB using 20ml 1.33% liposomal bupivacaine only (LB20-ACB) (Experimental): adductor canal block with 20ml 1.33% liposomal bupivacaine (266mg)
  Interventions: Drug: 1.33% liposomal bupivacaine only

INTERVENTIONS:
Drug: 0.5% standard bupivacaine only — 20ml 0.5% standard bupivacaine only
  Arms: ACB using 20ml 0.5% standard bupivacaine (SB-ACB)
Drug: 1.33% liposomal bupivacaine with 0.5% standard bupivacaine — 10ml 1.33% liposomal bupivacaine (133mg) plus 10ml 0.5% standard bupivacaine
  Arms: ACB using 10ml 1.33% liposomal bupivacaine with 10 ml 0.5% standard bupivacaine (LB10-ACB)
Drug: 1.33% liposomal bupivacaine only — 20ml 1.33% liposomal bupivacaine (266mg)
  Arms: ACB using 20ml 1.33% liposomal bupivacaine only (LB20-ACB)

SUMMARY:
Total knee arthroplasty is a commonly performed orthopaedic surgery for the treatment of end-stage osteoarthritis when conservative management becomes ineffective. TKA is associated with significant acute postoperative pain and many patients experience severe postoperative pain despite the use of multimodal analgesia. Poor acute postoperative pain control impacts rehabilitation, prolongs recovery and increases opioid consumption and chronic post-surgical pain.

Liposomal bupivacaine (Exparel, Pacira Pharmaceuticals Inc, Parsippany, New Jersey, USA) is a multivesicular formulation of bupivacaine that prolongs drug release and can extend the duration of analgesia. The adductor canal block (ACB) has been shown to reduce pain intensity and opioid consumption after total knee arthroplasty. The use of liposomal bupivacaine in the adductor canal block has recently been FDA-approved. However, the results of its efficacy from existing clinical trials have been mixed. In addition, the doses in the clinical trials have been different, and the optimal dose for perineural application of liposomal bupivacaine is unclear, including for the adductor canal block.

In this project, the investigators propose to conduct a randomized controlled trial to investigate the effect of different doses of liposomal bupivacaine in the adductor canal block on acute postoperative pain intensity and opioid consumption after robotic assisted total knee arthroplasty. The investigators will also assess secondary outcomes including knee functional scores, chronic pain and quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80 years old
* Scheduled for elective primary unilateral total knee arthroplasty (TKA) with robotic surgery
* Able to speak and understand Cantonese or Mandarin or English
* Able to provide informed oral and written consent

Exclusion Criteria:

* Revision TKA
* Single-stage bilateral TKA
* Complex primary TKA requiring use of stem/augment/constrained liner
* Surgeries with significant intraoperative complications which may alter rehabilitation protocol eg collateral ligament injury, fracture requiring fixation
* Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors
* History of chronic pain other than chronic knee pain
* History of immunosuppression
* Chronic use of glucocorticoids
* Chronic opioid use (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* History of congestive heart failure (NYHA 2)
* Alcohol or drug abuse
* Impaired renal function (defined as effective glomerular filtration rate < 30ml/min/1.73m2
* Impaired liver function (defined as plasma bilirubin over 34mol/L; international normalized ratio [INR] >= 1.7, alanine aminotransferase [ALT] over 100U/L, aspartate aminotransferase [AST] over 100U/L)
* Coagulopathy (platelet count <100,000/ml and/or INR >= 1.5) or the use of anticoagulants (not including aspirin) that precludes the use of adductor canal blocks
* Pre-existing neurological or muscular disorders
* Psychiatric illness
* Impaired mental state
* Pregnancy
* Local infection
* On immunosuppressants
* High body mass index (BMI) (>=40)
* Patient refusal for regional nerve blocks or to conduct clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Weighted area under curve (AUC) pain score | The first 48 hours after surgery when the patient is at rest
  Pain severity would be rated at rest after surgery using numerical rating scale (NRS) with 0 to 10 where 0=no pain and 10=the worst possible pain

SECONDARY OUTCOMES:
NRS pain scores | from after surgery to postoperative day 7
  NRS pain scores at rest and with movement (active knee flexion) from after surgery to postoperative day (POD) 7, ranging 0-10, with higher scores indicating more severe pain.
Oxynorm consumption | Postoperative day 1-7
  Oxynorm consumption from postoperative day (POD) 1-7
Overall Benefit of Analgesic Score (OBAS) | Postoperative day (POD) 1-7
  Overall Benefit of Analgesic Score (OBAS) from postoperative day (POD) 1-7 (range, 0 [best] to 28 [worst])
Plasma level of bupivacaine and ropivacaine | Blood will be collected during induction, at 12 hours, 24 hours, 48 hours, and 72 hours after ACB.
  Plasma level of bupivacaine and ropivacaine before and after surgery
Quality of Recovery Questionnaire (QoR-9) | Postoperative day 1
  Quality of Recovery Questionnaire (QoR-9) on postoperative day 1, ranging from 0 to 18, with higher scores indicating good recovery after anaesthesia.
Rehabilitation parameters (range of maximal active knee flexion) | While the patient is in hospital from postoperative day 0, day 1, and day 2.
  Range of maximal active knee flexion will be assessed by the physiotherapists while the patient is in hospital.
Rehabilitation parameters (quadricep power) | While the patient is in hospital from postoperative day 0, day 1, and day 2.
  Quadricep power will be assessed by the physiotherapists while the patient is in hospital.
  Ratings:
  0 - no muscle contraction
  1. - Move w/o gravity
  2. - Raise then drop down immediately
  3. - Raise against gravity w/o resistance
  4. - Raise against gravity w/some resistance
  5. - Raise against gravity w/ full resistance
Rehabilitation parameters (ability to perform straight leg raising) | While the patient is in hospital from postoperative day 0, day 1, and day 2.
  Ability to perform straight leg raising will be assessed by the physiotherapists while the patient is in hospital. Ratings (Yes/ No).
Rehabilitation parameters (walking distance) | While the patient is in hospital from postoperative day 0, day 1, and day 2.
  Walking distance (in metres) will be assessed by the physiotherapists while the patient is in hospital.
Rehabilitation parameters (Duration of hospital stay) | estimated on average of postoperative day 7 at the date of discharge from hospital
  No. of hospitalization days from admission to discharge
Rehabilitation parameters (discharge location) | estimated on average of postoperative day 7 at the date of discharge from hospital
  Home or rehabilitation center
Opioid-related side effects | While the patient is in hospital from postoperative day 0, 1, and 2.
  Presence or absence of pruritus, dizziness, nausea, and vomiting will be recorded.
Potential side effects related to adductor canal block (ACB) | While the patient is in hospital from postoperative day 0, 1, and 2.
  Presence or absence of local anaesthetic toxicity, neurological injury, and intravascular injection will be recorded.
Analgesic block duration | While the patient is in hospital at postoperative day 1
  Measured in time to return of pain (When did your pain relief from the block completely wear off?), time to sensory resolution (When did your numbness completely resolve and return to normal?), and time to motor resolution (When did your arm or hand weakness resolve and return to normal?)
Sensory and motor assessment | While the patient is in hospital from post-block 2 hours, 6 hours, 12 hours, and 24 hours.
  The affected lower limb will be measured.
  Sensory assessment (Sensation to pin prick), rating from 0 (no sensation) to 10 (normal sensation)
  Motor assessment
  * Straight leg raising achieved Ratings (Yes/ No)
  * Quadriceps power
  Ratings:
  0 - no muscle contraction
  1. - Move w/o gravity
  2. - Raise then drop down immediately
  3. - Raise against gravity w/o resistance
  4. - Raise against gravity w/some resistance
  5. - Raise against gravity w/ full resistance
quality of life (SF12v2) | at 6 weeks and at 3 and 6 months after surgery
  Eight domains of SF-12v2 (HK) are measured on a scale ranging from 0 to 100. A higher domain score indicates a better HRQoL.
Identification Pain Questionnaire for Neuropathic Pain (ID-NeP) | at 6 weeks, 3 months and 6 months postoperatively
  Neuropathic pain will be assessed using Identification Pain Questionnaire for Neuropathic Pain (ID-NeP), consisting of six items: "Yes" answers to questions 1-5 were given a score of 1, while "yes" answer to question 6 scored -1. "No" answers to questions 1-5 were given a score of 0, while "yes" answer to question 6 scored 0.
Knee Society Knee Function Score | at 6 weeks, 3 months and 6 months postoperatively
  Knee Society Knee Function Score at 6 weeks, 3 months and 6 months postoperatively, from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Chronic post-surgical pain | at 6 weeks, 3 months and 6 months postoperatively
  The presence or absence of chronic post-surgical pain, pain scores if present.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Result] Culliton SE, Bryant DM, MacDonald SJ, Hibbert KM, Chesworth BM. Validity and Internal Consistency of the New Knee Society Knee Scoring System. Clin Orthop Relat Res. 2018 Jan;476(1):77-84. doi: 10.1007/s11999.0000000000000014. PMID 29529620
- [Result] Portenoy R. Development and testing of a neuropathic pain screening questionnaire: ID Pain. Curr Med Res Opin. 2006 Aug;22(8):1555-65. doi: 10.1185/030079906X115702. PMID 16870080
- [Result] Chan MT, Lo CC, Lok CK, Chan TW, Choi KC, Gin T. Psychometric testing of the Chinese quality of recovery score. Anesth Analg. 2008 Oct;107(4):1189-95. doi: 10.1213/ane.0b013e318184b94e. PMID 18806027
- [Result] Lam ET, Lam CL, Fong DY, Huang WW. Is the SF-12 version 2 Health Survey a valid and equivalent substitute for the SF-36 version 2 Health Survey for the Chinese? J Eval Clin Pract. 2013 Feb;19(1):200-8. doi: 10.1111/j.1365-2753.2011.01800.x. Epub 2011 Nov 29. PMID 22128754
- [Result] Lehmann N, Joshi GP, Dirkmann D, Weiss M, Gulur P, Peters J, Eikermann M. Development and longitudinal validation of the overall benefit of analgesia score: a simple multi-dimensional quality assessment instrument. Br J Anaesth. 2010 Oct;105(4):511-8. doi: 10.1093/bja/aeq186. Epub 2010 Aug 6. PMID 20693179
- [Result] Cohen, J., Statistical power analysis for the behavioral sciences. 2013: routledge.
- [Result] Quaye A, McAllister B, Garcia JR, Nohr O, Laduzenski SJ, Mack L, Kerr CR, Kerr DA, Razafindralay CN, Richard JM, Craig WY, Rodrigue S. A prospective, randomized trial of liposomal bupivacaine compared to conventional bupivacaine on pain control and postoperative opioid use in adults receiving adductor canal blocks for total knee arthroplasty. Arthroplasty. 2024 Feb 1;6(1):6. doi: 10.1186/s42836-023-00226-y. PMID 38297390
- [Result] Malige A, Pellegrino AN, Kunkle K, Konopitski AK, Brogle PJ, Nwachuku CO. Liposomal Bupivacaine in Adductor Canal Blocks Before Total Knee Arthroplasty Leads to Improved Postoperative Outcomes: A Randomized Controlled Trial. J Arthroplasty. 2022 Aug;37(8):1549-1556. doi: 10.1016/j.arth.2022.03.073. Epub 2022 Mar 26. PMID 35351553
- [Result] Hungerford M, Neubauer P, Ciotola J, Littleton K, Boner A, Chang L. Liposomal Bupivacaine vs Ropivacaine for Adductor Canal Blocks in Total Knee Arthroplasty: A Prospective Randomized Trial. J Arthroplasty. 2021 Dec;36(12):3915-3921. doi: 10.1016/j.arth.2021.08.017. Epub 2021 Aug 21. PMID 34556382
- [Result] Hubler CP, Bevil KM, Greiner JJ, Hetzel SJ, Borden SB, Cios HA. Liposomal Bupivacaine Versus Standard Bupivacaine in the Adductor Canal for Total Knee Arthroplasty: A Randomized, Controlled Trial. Orthopedics. 2021 Jul-Aug;44(4):249-255. doi: 10.3928/01477447-20210621-01. Epub 2021 Jul 1. PMID 34292820
- [Result] Lv J, Huang C, Wang Z, Ou S. Adductor canal block combined with local infiltration analgesia versus isolated adductor canal block in reducing pain and opioid consumption after total knee arthroplasty: a systematic review and meta-analysis. J Int Med Res. 2020 Aug;48(8):300060520926075. doi: 10.1177/0300060520926075. PMID 32776794
- [Result] Li Y, Li A, Zhang Y. The efficacy of combined adductor canal block with local infiltration analgesia for pain control after total knee arthroplasty: A meta-analysis. Medicine (Baltimore). 2018 Dec;97(49):e13326. doi: 10.1097/MD.0000000000013326. PMID 30544393
- [Result] Zuo W, Guo W, Ma J, Cui W. Dose adductor canal block combined with local infiltration analgesia has a synergistic effect than adductor canal block alone in total knee arthroplasty: a meta-analysis and systematic review. J Orthop Surg Res. 2019 Apr 11;14(1):101. doi: 10.1186/s13018-019-1138-5. PMID 30971284
- [Result] Ilfeld BM, Eisenach JC, Gabriel RA. Clinical Effectiveness of Liposomal Bupivacaine Administered by Infiltration or Peripheral Nerve Block to Treat Postoperative Pain. Anesthesiology. 2021 Feb 1;134(2):283-344. doi: 10.1097/ALN.0000000000003630. PMID 33372949
- [Result] Jiang X, Wang QQ, Wu CA, Tian W. Analgesic Efficacy of Adductor Canal Block in Total Knee Arthroplasty: A Meta-analysis and Systematic Review. Orthop Surg. 2016 Aug;8(3):294-300. doi: 10.1111/os.12268. PMID 27627711
- [Result] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Result] Lavand'homme PM, Kehlet H, Rawal N, Joshi GP; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Pain management after total knee arthroplasty: PROcedure SPEcific Postoperative Pain ManagemenT recommendations. Eur J Anaesthesiol. 2022 Sep 1;39(9):743-757. doi: 10.1097/EJA.0000000000001691. Epub 2022 Jul 20. PMID 35852550